CLINICAL TRIAL: NCT02217917
Title: A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo Controlled, Single And Multiple Ascending Dose Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Rivipansel (pf 06460031) Following Subcutaneous Administration With Rhuph20 (pf 06744547) In Healthy Subjects
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous Rivipansel With rHuPH20 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: B5201007; 2014-002748-41 (EudraCT Number)
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: Healthy subjects; Randomized; Double-blind; Single ascending dose; Multiple ascending dose
MeSH Terms: interventions — rivipansel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Single ascending dose in 3 period cross-over design (with optional 4th period)
  Interventions: Drug: Rivipansel; Drug: Placebo
- Cohort 2 (Experimental): Multiple ascending dose
  Interventions: Drug: Rivipansel; Drug: Placebo
- Cohort 3 (Experimental): Multiple ascending dose
  Interventions: Drug: Rivipansel; Drug: Placebo

INTERVENTIONS:
Drug: Rivipansel — Rivipansel administered as a single dose subcutaneously with rHuPH20 in cross-over fashion. Each subject may receive up to 4 study treatments (placebo and up to 3 doses of rivipansel). The planned dose levels are 350 mg, 1210 mg, and 4200 mg (these are subject to change based on emerging data).
  Arms: Cohort 1
Drug: Placebo — Matched Placebo administered as single dose subcutaneously with rHuPH20.
  Arms: Cohort 1
Drug: Rivipansel — Rivipansel administered q12h for 7 days (a total of 13 doses) subcutaneously with rHuPH20. Planned doses are 1400 mg loading and 700 mg maintenance for 12 doses (these are subject to change based on emerging data).
  Arms: Cohort 2
Drug: Rivipansel — Rivipansel administered q12h for 7 days (a total of 13 doses) subcutaneously with rHuPH20. Planned doses are 2800 mg loading and 1400 mg maintenance for 12 doses (these are subject to change based on emerging data).
  Arms: Cohort 3
Drug: Placebo — Matched Placebo administered q12h for 7 days (a total of 13 doses) subcutaneously with rHuPH20.
  Arms: Cohort 2; Cohort 3

SUMMARY:
This is a 2 part study designed to provide an initial assessment on the safety, tolerability, and PK of rivipansel, following single ascending (Part 1) and multiple ascending dosing (Part 2) given subcutaneously with rHuPH20, in healthy subjects. Part 1 of the study will be conducted using a cross-over design while Part 2 of the study will be conducted using a parallel design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive.
* Body Mass Index 17.5 - 30.5 kg/m2 and body weight >50 kg at Screening.
* Normal skin without potentially obscuring features in the area intended for infusion.
* Subjects willing to defer receiving prophylactic immunizations (eg, influenza or pneumococcal vaccines) during the study.
* Evidence of a personally signed and dated informed consent document indicating that the subject or a legally acceptable representative has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of a recent major surgery (within 3 months of screening).
* Serious infection within 1 month of screening.
* Subjects with chronic skin condition that may interfere in the assessment of emergent safety data.
* A positive urine drug screen.
* Known sensitivity to hyaluronidases.
* History of hepatitis or positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibodies (HCV).
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) | Baseline up to 7 days of dosing
Assessment of cardiac conduction intervals as assessed via 12-lead electrocardiogram (ECG) | Baseline up to 7 days of dosing
Assessment of vital signs (including blood pressure and pulse rate) | Baseline up to 7 days of dosing
Assessment of clinical laboratory tests | Baseline up to 7 days of dosing

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Time to Reach Maximum Observed Plasma Concentration (Tmax) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Dose-Normalized Cmax for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Dose-Normalized AUClast for rivipansel | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Dose-Normalized AUCinf for rivipansel | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Plasma Decay Half-Life (t1/2) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Apparent Clearance (CL/F) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Apparent Volume of Distribution (Vz/F) for rivipansel following single dose | Samples are collected pre-dose and at 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72 H following single dose administration
Maximum Observed Plasma Concentration (Cmax) for rivipansel following multiple dose | Days 1, 7
Time to Reach Maximum Observed Plasma Concentration (Tmax) for rivipansel following multiple dose | Days 1, 7
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) for rivipansel following multiple dose administration, where tau is 12 hours | Days 1, 7
Dose-Normalized Cmax for rivipansel following multiple dose administration | Days 1, 7
Dose-Normalized AUCtau for rivipansel following multiple dose administration | Days 1, 7
Plasma Decay Half-Life (t1/2) for rivipansel following multiple dose | Day 7
Minimum Observed Plasma Concentration (Cmin) for rivipansel following multiple dose | Day 7
Apparent Clearance (CL/F) for rivipansel following multiple dose | Day 7
Peak to Trough Ratio (PTR) of plasma concentration for rivipanselmultiple dose administration | Day 7
Accumulation ratio for Area Under the Curve during the dosing interval (Rac) for rivipansel | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium